CLINICAL TRIAL: NCT03322930
Title: Rod Sensitivity in Age-related Macular Degeneration (AMD) and Retinitis Pigmentosa (RP)
Status: Completed | Type: Observational
Sponsor: Retina Foundation of the Southwest (Other)
Responsible Party: Sponsor
Other Study IDs: STU082017-084
Record Dates: First submitted 2017-10-24; First posted 2017-10-26 (Actual); Results first posted 2019-12-04 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Retinitis Pigmentosa; AMD
Keywords: microperimetry; rod visual fields
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retinitis Pigmentosa: patients with a diagnosis of retinitis pigmentosa and reduced rod function on baseline testing
  Interventions: Diagnostic Test: Rod sensitivity
- Age-related Macular Degeneration: patients with a diagnosis of intermediate AMD and reduced rod function on baseline testing
  Interventions: Diagnostic Test: Rod sensitivity

INTERVENTIONS:
Diagnostic Test: Rod sensitivity — diagnostic test for rod loss in central retina

SUMMARY:
A new fundus-guided microperimeter (MP-3S) has been developed by Nidek, Inc. to track the fundus of the patient and present stimuli in specific anatomically-defined locations. Furthermore, this tracking means that exactly the same locations can be tested on subsequent (follow-up) visits. The investigators will use a method called two-color perimetry to map rod and cone sensitivity on this device. With this technique, the sensitivity difference (blue-red) to chromatic test stimuli can be used to determine whether rods, cones or both photoreceptor systems mediate the threshold at a given location in the macula.

DETAILED DESCRIPTION:
Despite recent advances in understanding the pathogenesis of retinitis pigmentosa (RP) and age-related macular degeneration (AMD), precise characterization of the disease phenotype remains elusive. In both diseases, much of the focus has necessarily been on the loss of cone function, since visual fields, acuity and contrast sensitivity are typically measured under photopic conditions. In RP, we need a greater understanding of patterns of rod loss since most disease-causing mutations affect primarily rods. In AMD, recent findings have shown that scotopic sensitivity can be much more affected than conventional photopic measurements such as visual acuity. For patients, however, it is difficult to maintain stable fixation, especially when central vision is compromised. A new fundus-guided microperimeter, the MP-3S, has been developed by Nidek, Inc. to circumvent this problem. The investigators will evaluate the value of this device for following rod and cone loss in patients with either RP or AMD.

ELIGIBILITY:
Inclusion Criteria:

* clear media
* diagnosis of RP or non neovascular AMD
* normal volunteers

Exclusion Criteria:

* exudative AMD
* other eye diseases that could cause vision loss
* physical ailments that would preclude comfortable testing
* unable to provide informed consent

Ages: 10 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: 50 subjects with retinitis pigmentosa 50 patients with AMD 10 normal volunteers ages 18 to 40 and 10 normal volunteers ages over age 55 years
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Birch, PhD, Principal Investigator — Retina Foundation of the Southwest
Locations (1):
- Retina Foundation of the Southwest, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
anonymized rod visual fields

REFERENCES:
- See also: Retina Foundation of the Southwest website — http://retinafoundation.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: patients recruited from medical clinic (Texas Retina Associates)
Groups:
- Patients With a Diagnosis of Retinitis Pigmentosa: patients with a diagnosis of retinitis pigmentosa
  Rod sensitivity: diagnostic test for rod loss in central retina
- Patients With Intermediate Age-related Macular Degeneration: patients with a diagnosis of intermediate AMD
  Rod sensitivity: diagnostic test for rod loss in central retina
Period: Overall Study
Arm/Group | Patients With a Diagnosis of Retinitis Pigmentosa | Patients With Intermediate Age-related Macular Degeneration
Started (recruitment of 40 patients) | 20 (recruitment of 20 patients with retinitis pigmentosa) | 20 (recruitment of 20 patients with macular degeneration)
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Patients With a Diagnosis of Intermediate AMD: patients with a diagnosis of intermediate AMD
  Rod sensitivity: diagnostic test for rod loss in central retina
- Total: Total of all reporting groups
Arm/Group | Patients With a Diagnosis of Retinitis Pigmentosa | Patients With a Diagnosis of Intermediate AMD | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 5 | 25
  >=65 years | 0 | 15 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 15 | 27
  Male | 8 | 5 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 18 | 20 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 2 | 1 | 3
  White | 12 | 17 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Rod Sensitivity Within the Central Retina as Measured on the Nidek MP-3S
Description: Number of participants with rod sensitivity measured in decibels at multiple retinal locations within the central retina
Time Frame: through study completion, an average of 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With a Diagnosis of Retinitis Pigmentosa | Patients With a Diagnosis of Intermediate AMD
Number analyzed (Participants) | 20 | 20
Participants | 7 | 20
Statistical Analysis 1: Comparison: Patients With a Diagnosis of Retinitis Pigmentosa vs Patients With a Diagnosis of Intermediate AMD; Test type: Other; p < 0.05, t-test, 2 sided — calculated from data; mean sensitivity for group; Coefficient of Repeatability for multiple tests per patient

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Patients With a Diagnosis of Retinitis Pigmentosa | Patients With a Diagnosis of Intermediate AMD
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-10-24): https://cdn.clinicaltrials.gov/large-docs/30/NCT03322930/Prot_000.pdf